CLINICAL TRIAL: NCT00809276
Title: Trial of Allogeneic BMT for Hematologic Malignancies Using HLA-matched Related or Unrelated Donors With Fludarabine and IV Busulfan as Pre-transplant Conditioning Followed by Post-transplant Immunosuppression With High-dose Cyclophosphamide
Brief Title: Allo BMT Using Matched Related/Unrelated Donors With FluBu and HiCY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Fred Hutchinson Cancer Center (Other); Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0844; NA_00017193 (Other: JHMIRB)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Lymphoma; Multiple Myeloma; Leukemia; Myelodysplastic Syndrome
Keywords: Acute lymphocytic leukemia (ALL); Acute myeloid leukemia (AML); Acute Leukemia; Refractory or Relapsed AML; Myelodysplastic syndrome (MDS); Chronic myeloid leukemia (CML); Chronic myelomonocytic leukemia; Hodgkin's Lymphoma; Non-Hodgkin's lymphoma; Philadelphia-negative myeloproliferative disorder; Hematologic Malignancies; Transplantation; Busulfan; Fludarabine; Cytoxan; Bone Marrow; Allogeneic; Related donor; unrelated donor
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Hodgkin Disease; Lymphoma, Non-Hodgkin; Hematologic Neoplasms | interventions — Busulfan; fludarabine; Cyclophosphamide; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Busulfan, Fludarabine, Cytoxan — Busulfan once a day for 4 days
  Fludarabine once a day for 4 days
  Bone marrow transplant
  Cytoxan two doses
  Other Names: BMT; Cyclophosphamide; Allogeneic; Transplantation

SUMMARY:
The purpose of this research is to find the most effective and least toxic way to prevent GVHD after BMT.

DETAILED DESCRIPTION:
A person who has cancer of the blood or lymph glands can be treated by bone marrow transplantation (BMT). BMT has developed over several decades of research on both animal and human subjects as an effective treatment of various malignant and nonmalignant hematologic diseases. Many hematologic malignancies can be successfully treated with a combination of high-dose chemotherapy or chemo-radiotherapy and transplantation of allogeneic bone marrow or peripheral blood stem cells (alloBMT)

However, a possible side effect of BMT is graft versus host disease (GVHD). GVHD occurs when cells of the donor's immune system, which are present in the bone marrow, attack the BMT recipient's normal tissue. Prevention of GVHD is important for the success of the bone marrow transplant. This research is being done to find the most effective and least toxic way to prevent GVHD after BMT

ELIGIBILITY:
Inclusion Criteria:

* Patients ages between 0 to and 65 years of age.
* Patient must have a genotypically HLA-identical sibling, a phenotypically matched first-degree relative or an unrelated matched donor.
* Acute lymphocytic leukemia (ALL) in CR1 with high risk features
* Acute myeloid leukemia (AML) in CR1 with high risk features defined as:

  i. Greater than 1 cycle of induction therapy required to achieve remission, ii. Preceding myelodysplastic syndrome (MDS) other than myelofibrosis, secondary AML iii. Presence of Flt3 mutations or internal tandem duplications, iv. FAB M6 or M7 classification or adverse cytogenetics for overall survival such as those associated with MDS, M6, M7 leukemia, or v. Complex karyotype [> 3 abnormalities]
* Acute Leukemias in 2nd or greater remission
* Refractory or Relapsed AML
* AML transformed from MDS
* Myelodysplastic syndrome (MDS) beyond refractory anemia
* Chronic myeloid leukemia (CML)
* Chronic myelomonocytic leukemia
* Philadelphia-negative myeloproliferative disorder
* Relapsed chemotherapy-sensitive Hodgkin's or Non-Hodgkin's lymphoma
* Multiple Myeloma-Stage III

Exclusion Criteria:

* Prior autologous or allogeneic stem cell transplant.
* Performance status greater than 2
* Active infection.
* Inadequate cardiac function; arrythmias or symptomatic cardiac disease.
* Inadequate pulmonary function; FEV1, FVC, DLCO <50% of predicted
* Inadequate Serum creatinine clearance <60
* InadequatebHepatic function
* Positive serology for HIV-1, 2 or HTLV-1, 2.
* Pregnancy. Female patient must have negative pregnancy test

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Luznik, MD, Study Chair — Johns Hopkins University
Locations (3):
- United States (3):
  - The Sydney Kimmel Comprehensive Cancer center, Baltimore, Maryland
  - Marcos deLima, MD, Houston, Texas
  - Paul V. O'Donnell, M.D., Ph.D., Seattle, Washington

REFERENCES:
- [Derived] Kanakry CG, O'Donnell PV, Furlong T, de Lima MJ, Wei W, Medeot M, Mielcarek M, Champlin RE, Jones RJ, Thall PF, Andersson BS, Luznik L. Multi-institutional study of post-transplantation cyclophosphamide as single-agent graft-versus-host disease prophylaxis after allogeneic bone marrow transplantation using myeloablative busulfan and fludarabine conditioning. J Clin Oncol. 2014 Nov 1;32(31):3497-505. doi: 10.1200/JCO.2013.54.0625. Epub 2014 Sep 29. PMID 25267759

RESULTS

PARTICIPANT FLOW:
Groups:
- BuFlu Transplant: Myeloablative bone marrow transplant with busulfan and fludarabine conditioning Post-transplantation cyclophosphamide as single-agent graft-versus-host-disease prophylaxis
Period: Overall Study
Arm/Group | BuFlu Transplant
Started | 92
Completed | 92
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BuFlu Transplant
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 49 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Optimal Regimen of Post-graft Immunosuppression With High-dose Cy Following Fludarabine, Busulfan, and Transplantation of Fully HLA-matched Bone Marrow That Leads to an Acceptable Incidence of Grades III/IV Acute GVHD
Description: Percentage of participants with grade III-IV acute graft versus host disease (GVHD). GVHD is graded on a combination of skin symptoms (rash), gut symptoms (diarrhea), and liver symptoms (using a lab test called bilirubin). Grades range from I to IV, where I is the least severe and IV is the most severe.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BuFlu Transplant
Number analyzed (Participants) | 92
percentage of participants | 15 [8 to 23]

ADVERSE EVENTS:
Time Frame: Up to 100 days after bone marrow transplant.
Description: Systematically monitored through at least Day 60.
Arm/Group | BuFlu Transplant
Serious Adverse Events (participants affected / at risk) | 40/92
Other Adverse Events (participants affected / at risk) | 34/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BuFlu Transplant (N=92)
Primary graft failure (Blood and lymphatic system disorders) | 5
Death (Investigations) | 8
ALT elevation grade 3-4 (Investigations) | 8
AST elevation grade 3-4 (Investigations) | 6
Hyperbilirubinemia grade 3-4 (Investigations) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Alkaline phosphatase elevated grade 3-4 (Investigations) | 3
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Gastritis and ileitis (Gastrointestinal disorders) | 1
Hemorrhagic cystitis (Renal and urinary disorders) | 2
Hyperuricemia (Investigations) | 1
Hypokalemia (Investigations) | 1
Hypotension (Cardiac disorders) | 1
Infection (Infections and infestations) | 12
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Mucositis (Gastrointestinal disorders) | 19
Neutropenic fever (Infections and infestations) | 11
Rash (Skin and subcutaneous tissue disorders) | 1
Renal toxicity (Renal and urinary disorders) | 1
Subdural hematoma (Blood and lymphatic system disorders) | 1
Secondary graft failure (Blood and lymphatic system disorders) | 2
Diffuse alveolar hemorrhage (Blood and lymphatic system disorders) | 1
Idiopathic pulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BuFlu Transplant (N=92)
AST elevation grade 3-4 (Investigations) | 11
ALT elevation grade 3-4 (Investigations) | 20
Mucositis (Gastrointestinal disorders) | 6
Engraftment > Day 28 (Investigations) | 11
Hyperbilirubinemia grade 3-4 (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No